CLINICAL TRIAL: NCT02546323
Title: A Randomized, Double-blind, Placebo-controlled, Multicenter Parallel Group Phase 3 Study Measuring the Effect of Rosuvastatin 20 mg on Carotid Intima-Media Thickness in Chinese Subjects
Brief Title: A phase3 Study Measuring the Effect of Rosuvastatin 20 mg on Carotid Intima-Media Thickness in Chinese Subjects With Subclinical Atherosclerosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D3565C00003
Record Dates: First submitted 2015-08-26; First posted 2015-09-10 (Estimated); Results first posted 2019-12-11 (Actual); Last update posted 2019-12-11 (Actual); Status verified 2019-10

CONDITIONS: Atherosclerosis
Keywords: Rosuvastatin 20 mg treatment, Carotid Intima-Media Thickness, Chinese subjects, Subclinical atherosclerosis
MeSH Terms: conditions — Atherosclerosis | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rosuvastatin (Experimental): 20 mg tablets, Daily oral dose
  Interventions: Drug: Rosuvastatin
- Placebo (Placebo Comparator): Matching placebo tablets
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rosuvastatin — 20mg tablets, orally once daily for the duration of the 104-week treatment period
  Other Names: Crestor
  Arms: Rosuvastatin
Drug: Placebo — Matching placebo tablets, orally once daily for the duration of the 104-week treatment period.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the effects of of rosuvastatin 20 mg compared to placebo for treating Chinese patients with subclinical atherosclerosis.

DETAILED DESCRIPTION:
This study is a randomized, double-blind, placebo-controlled, multicenter parallel group study assessing the effects of rosuvastatin 20 mg treatment for 104 weeks on the change in intimamedia thickness (IMT) of the common carotid artery (CCA), carotid bulb, and internal carotid artery (ICA) in adult Chinese subjects with subclinical atherosclerosis.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent prior to any study-specific procedures
* Male aged ≥45 and <70 years or female aged ≥55 and <70 years
* Subjects with only hypertension (as defined blood pressure ≥140/90 mmHg or on antihypertensive treatment) and age as CVD risk factors and subjects without hypertension who have 3 or more other risk factors (including age) must have "Fasting LDL C of ≥120 mg/dL (3.1 mmol/L) and <160 mg/dL (4.1mmol/L)"; Subjects without hypertension who have fewer than 3 other risk factors (including age) must have "Fasting LDL-C of ≥120 mg/dL (3.1 mmol/L) and <190 mg/dL (4.9 mmol/L)"
* Triglycerides <500 mg/dL (5.65 mmol/L) at Visit 1
* HDL-C levels ≤60 mg/dL (1.6 mmol/L) at Visit 1
* Maximum IMT ≥1.2 mm and <3.5 mm at any location in the carotid ultrasound scans conducted at both Visit 2 and Visit 3
* Willing to follow all study procedures including study visits, fasting blood draws, and compliance with study treatment regimen

Exclusion Criteria:

* Use of pharmacologic lipid-lowering medications (eg, statins, fibrate derivatives,bile acid binding resins, niacin, or its analogues at doses >400 mg or prescribed Chinese traditional drugs), including cholesterol-absorption inhibitors (CAIs), and CAI/statin combination, within 12 months prior to Visit 1
* Current or recent (within 2 weeks of Visit 1) use of supplements known to alter lipid metabolism (eg, soluble fibers [including >2 teaspoons Metamucil® or psyllium-containing supplement per day] or other dietary fiber supplements, marine oils, sterol/stanol products, or other supplement determined at the discretion of the investigator)
* History of hypersensitivity reactions to other HMG-CoA reductase inhibitors
* Pregnant women, women who are breast-feeding, and women of childbearing potential who are not using chemical or mechanical contraception or who have a positive serum pregnancy test
* Clinical evidence of coronary artery disease (CAD) or any other atherosclerotic disease such as angina, MI, transient ischemic attack, symptomatic CAD, cerebrovascular accident, percutaneous coronary intervention, coronary artery bypass graft, peripheral arterial disease, abdominal aortic aneurysm
* History of cancer (other than basal cell carcinoma) in the past 2 years
* Uncontrolled hypertension defined as either a mean resting diastolic blood pressure of ≥110 mmHg or a resting systolic blood pressure of ≥180 mmHg recorded at any time during the screening period
* History of diabetes mellitus or current diabetes mellitus
* Uncontrolled hypothyroidism defined as a thyroid stimulating hormone (TSH) >1.5 times the upper limit of normal (ULN) at Visit 1 or subjects whose thyroid replacement therapy was initiated within the last 3 months
* History of heterozygous or homozygous familial hypercholesterolemia or known hyperlipoproteinemia Types I, III, IV, or V (familial dysbetalipoproteinemia)
* Use of the disallowed concomitant medications within 12 months prior to Visit 1
* History of alcohol and/or drug abuse within the past 5 years
* Active liver disease or hepatic dysfunction as defined by elevations of ≥1.5 x ULN at Visit 1 in any of the following liver function tests: ALT, AST or bilirubin
* Serum creatine kinase (CK) >3 x ULN at Visit 1
* Serum creatinine >2.0 mg/dL (177 mmol/L) recorded during the screening period
* Participation in another investigational drug study, and having ingested investigational drug ≤4 weeks before enrollment in the screening period
* Previous randomization in the present study
* History of a significant medical or psychological condition that, in the opinion of the investigator, would compromise the subject's safety or successful participation in the study
* Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site)

Ages: 45 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 543 (Actual)
Dates: Start 2015-09-17 (Actual); Primary Completion 2019-01-29 (Actual); Study Completion 2019-01-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yongjun Wang, M.D., Principal Investigator — Beijing Tian Tan Hospital, Capital Medical University; Yundai Chen, M.D., Principal Investigator — Chinese PLA General Hospital
Locations (15):
- China (15):
  - Research Site, Beijing
  - Research Site, Bengbu
  - Research Site, Changsha
  - Research Site, Chongqin
  - Research Site, Guangzhou
  - Research Site, Haerbin
  - Research Site, Nanchang
  - Research Site, Nanjing
  - Research Site, Ningbo
  - Research Site, Shanghai
  - Research Site, Shenyang
  - Research Site, Tianjin
  - Research Site, Wenzhou
  - Research Site, Wuhan
  - Research Site, Xi'an

REFERENCES:
- [Derived] Clezar CN, Flumignan CD, Cassola N, Nakano LC, Trevisani VF, Flumignan RL. Pharmacological interventions for asymptomatic carotid stenosis. Cochrane Database Syst Rev. 2023 Aug 4;8(8):CD013573. doi: 10.1002/14651858.CD013573.pub2. PMID 37565307
- [Derived] Zheng H, Li H, Wang Y, Li Z, Hu B, Li X, Fu L, Hu H, Nie Z, Zhao B, Wei D, Karlson BW, Bots ML, Meng X, Chen Y, Wang Y; METEOR-China Investigators. Rosuvastatin Slows Progression of Carotid Intima-Media Thickness: The METEOR-China Randomized Controlled Study. Stroke. 2022 Oct;53(10):3004-3013. doi: 10.1161/STROKEAHA.120.031877. Epub 2022 Aug 26. PMID 36017704
- [Derived] Wang Y, Wang A, Li H, Li Z, Hu B, Li X, Zheng H, Fu L, Hu H, Nie Z, Qin Y, Zhao B, Wei D, Karlson BW, Bots ML, Chen Y, Wang Y. Measuring effects on intima-media thickness: an evaluation of rosuvastatin in Chinese subjects with subclinical atherosclerosis-design, rationale, and methodology of the METEOR-China study. Trials. 2020 Nov 11;21(1):921. doi: 10.1186/s13063-020-04741-0. PMID 33176842
- See also: redacted protocol — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D3565C00003&attachmentIdentifier=d2d6e1c4-2f54-4e4f-a110-cba7a24b341c&fileName=D3565c00003_CSP_Redacted.pdf&versionIdentifier=
- See also: SAP_redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D3565C00003&attachmentIdentifier=6d21d378-0561-421c-88fb-99dc030ad2e8&fileName=D3565c00003_SAP_Redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Chinese patients with subclinical atherosclerosis and a 10-year ischemic cardiovascular disease (ICVD) risk of less than 10% (as assessed by the 2007 China Adult Dyslipidema Management Guidelines) were enrolled at 25 sites in China between 17 September 2015 and 29 January 2019.
Pre-assignment Details: Eligible patients with carotid intima-media thickness (CIMT) measurements of maximum CIMT ≥1.2 millimeters (mm) and <3.5 mm were randomized to receive either rosuvastatin 20 milligrams (mg) or corresponding placebo once daily. Randomization was stratified by ICVD risk (<5% or 5% to 10%).
Groups:
- Rosuvastatin 20 mg: Rosuvastatin 20 mg was administered in oral tablet form, once daily, for a 104-week (2-year) treatment period.
- Placebo: Placebo was administered in oral tablet form, once daily, for a 104-week (2-year) treatment period.
Period: Overall Study
Arm/Group | Rosuvastatin 20 mg | Placebo
Started (Randomized patients) | 272 | 271
Received Treatment | 272 | 268
Completed | 212 | 205
Not Completed | 60 | 66
Not completed — Withdrawal by Subject | 36 | 33
Not completed — Eligibility Criteria not Fulfilled | 0 | 1
Not completed — Adverse Event | 17 | 11
Not completed — Patient Specific Reasons | 1 | 2
Not completed — Lost to Follow-up | 2 | 3
Not completed — Non-compliance with Study Drug | 2 | 2
Not completed — Met Withdrawal Criteria | 2 | 14

BASELINE CHARACTERISTICS:
Population: The intent-to-treat (ITT) analysis set consisted of all randomized patients.
Groups:
- Total: Total of all reporting groups
Arm/Group | Rosuvastatin 20 mg | Placebo | Total
Number analyzed (Participants) | 272 | 271 | 543
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.0 (5.23) | 59.7 (4.96) | 59.4 (5.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 146 | 158 | 304
  Male | 126 | 113 | 239
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 272 | 271 | 543
10-year ICVD Risk [Count of Participants; unit: Participants] — ICVD risk as collected by the Interactive Voice/Web Response System.
  Participants
    <5% | 196 | 195 | 391
    ≥5% - <10% | 76 | 76 | 152

OUTCOME MEASURES:

1. Primary Outcome: Annualized Rate of Change in Mean of the Maximum (MeanMax) CIMT Measurements From Each of the 12 Carotid Artery Sites Based on All Scans Performed During the 104-Week Study Period
Description: CIMT measurements were made from ultrasound images of the common carotid artery (CCA), carotid bulb and internal carotid artery (ICA). The thickness of the intima and media was determined as the distance from the interface between the vessel lumen and the intima, to the interface between the media and the adventitia. Twelve carotid artery sites were scanned at each visit and the 3 images recorded at the 3 interrogation angles were measured to determine the maximum of the CIMT for a specific segment. The annualized rate of change in the MeanMax CIMT measurements from each of the 12 sites, based on all scans performed during the study, was determined using a multi-level linear mixed effects regression model that estimated mean annualized rate of change (mm/year) over the 104-week study period. The model fitted regression lines to profiles of CIMT values consisting of 2 pre-randomization values, 3 values from visits during the treatment period, and 2 end-of-study visits.
Time Frame: From baseline (pre-randomization Week -2 and Week -4) to end-of-study (Week 104).
Population: The ITT analysis set consisted of all randomized patients. Patients were analyzed according to the treatment to which they were randomized.
Measure: Mean (Standard Error); unit: mm/year
Arm/Group | Rosuvastatin 20 mg | Placebo
Number analyzed (Participants) | 272 | 271
mm/year | 0.0038 (0.00312) | 0.0142 (0.00317)
Statistical Analysis 1: Comparison: Rosuvastatin 20 mg vs Placebo; Comparison of annualized rate of change in MeanMax CIMT measurement difference between rosuvastatin 20 mg and placebo; Test type: Other; p = 0.020, Multi-level mixed effects model — Statistical significance of the MeanMax CIMT annualized rate of change between rosuvastatin 20 mg and placebo was evaluated using time-by-treatment interaction term in the model; Estimated mean difference = -0.0103, 95% CI 2-sided [-0.0191 to -0.0016], Standard Error of Mean 0.00445 — Randomized treatment group, time, time-by-treatment interaction, ICVD risk stratification, carotid artery site, center, age, sex, and scan reader were fixed effects. Random effects were the intercept and slope for individual patients

2. Secondary Outcome: Annualized Rate of Change in the MeanMax CIMT of the Near and Far Walls of the Right and Left CCA
Description: CIMT measurements were made from ultrasound images of the near and far walls of the right and left CCA. The thickness of the intima and media was determined as the distance from the interface between the vessel lumen and the intima, to the interface between the media and the adventitia. The 3 images recorded at the 3 interrogation angles were measured to determine the maximum of the CIMT for this segment. The annualized rate of change in the MeanMax CIMT measurements, based on all scans performed during the study, was determined using a multi-level linear mixed effects regression model that estimated mean annualized rate of change (mm/year) over the 104-week study period. The model fitted regression lines to profiles of CIMT values consisting of 2 pre-randomization values, 3 values from visits during the treatment period, and 2 end-of-study visits.
Time Frame: From baseline (pre-randomization Week -2 and Week -4) to end-of-study (Week 104).
Population: as for outcome 1
Measure: Mean (Standard Error); unit: mm/year
Arm/Group | Rosuvastatin 20 mg | Placebo
Number analyzed (Participants) | 272 | 271
mm/year | -0.0031 (0.00310) | 0.0079 (0.00315)
Statistical Analysis 1: Comparison: Rosuvastatin 20 mg vs Placebo; Comparison of annualized rate of change in MeanMax CIMT measurement difference between rosuvastatin 20 mg and placebo; Test type: Other; p = 0.013, Multi-level mixed effects model — [p-value comment as in outcome 1, analysis 1]; Estimated mean difference = -0.0110, 95% CI 2-sided [-0.0197 to -0.0024], Standard Error of Mean 0.00442 — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Annualized Rate of Change in the MeanMax CIMT of the Near and Far Walls of the Right and Left Carotid Bulb
Description: CIMT measurements were made from ultrasound images of the near and far walls of the right and left carotid bulb. The thickness of the intima and media was determined as the distance from the interface between the vessel lumen and the intima, to the interface between the media and the adventitia. The 3 images recorded at the 3 interrogation angles were measured to determine the maximum of the CIMT for this segment. The annualized rate of change in the MeanMax CIMT measurements, based on all scans performed during the study, was determined using a multi-level linear mixed effects regression model that estimated mean annualized rate of change (mm/year) over the 104-week study period. The model fitted regression lines to profiles of CIMT values consisting of 2 pre-randomization values, 3 values from visits during the treatment period, and 2 end-of-study visits.
Time Frame: From baseline (pre-randomization Week -2 and Week -4) to end-of-study (Week 104).
Population: as for outcome 1
Measure: Mean (Standard Error); unit: mm/year
Arm/Group | Rosuvastatin 20 mg | Placebo
Number analyzed (Participants) | 272 | 271
mm/year | 0.0067 (0.00634) | 0.0228 (0.00643)
Statistical Analysis 1: Comparison: Rosuvastatin 20 mg vs Placebo; Comparison of annualized rate of change in MeanMax CIMT measurement difference between rosuvastatin 20 mg and placebo; Test type: Other; p = 0.073, Multi-level mixed effects model — [p-value comment as in outcome 1, analysis 1]; Estimated mean difference = -0.0162, 95% CI 2-sided [-0.0339 to 0.0015], Standard Error of Mean 0.00903 — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Annualized Rate of Change in the MeanMax CIMT of the Near and Far Walls of the Right and Left ICA
Description: CIMT measurements were made from ultrasound images of the near and far walls of the right and left ICA. The thickness of the intima and media was determined as the distance from the interface between the vessel lumen and the intima, to the interface between the media and the adventitia. The 3 images recorded at the 3 interrogation angles were measured to determine the maximum of the CIMT for this segment. The annualized rate of change in the MeanMax CIMT measurements, based on all scans performed during the study, was determined using a multi-level mixed effects regression model that estimated mean annualized rate of change (mm/year) over the 104-week study period. The model fitted regression lines to profiles of CIMT values consisting of 2 pre-randomization values, 3 values from visits during the treatment period, and 2 end-of-study visits.
Time Frame: From baseline (pre-randomization Week -2 and Week -4) to end-of-study (Week 104).
Population: as for outcome 1
Measure: Mean (Standard Error); unit: mm/year
Arm/Group | Rosuvastatin 20 mg | Placebo
Number analyzed (Participants) | 272 | 271
mm/year | 0.0077 (0.00502) | 0.0120 (0.00511)
Statistical Analysis 1: Comparison: Rosuvastatin 20 mg vs Placebo; Comparison of annualized rate of change in MeanMax CIMT measurement difference between rosuvastatin 20 mg and placebo; Test type: Other; p = 0.547, Multi-level mixed effects model — [p-value comment as in outcome 1, analysis 1]; Estimated mean difference = -0.0043, 95% CI 2-sided [-0.0183 to 0.0097], Standard Error of Mean 0.00716 — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: Annualized Rate of Change in the Mean of the Mean (MeanMean) CIMT of the Near and Far Walls of the Right and Left CCA
Description: CIMT measurements were made from ultrasound images of the near and far walls of the right and left CCA. The thickness of the intima and media was determined as the distance from the interface between the vessel lumen and the intima, to the interface between the media and the adventitia. The 3 images recorded at the 3 interrogation angles were measured to determine the mean of the CIMT for this segment. The annualized rate of change in the MeanMean CIMT measurements, based on all scans performed during the study, was determined using a multi-level mixed effects regression model that estimated mean annualized rate of change (mm/year) over the 104-week study period. The model fitted regression lines to profiles of CIMT values consisting of 2 pre-randomization values, 3 values from visits during the treatment period, and 2 end-of-study visits.
Time Frame: From baseline (pre-randomization Week -2 and Week -4) to end-of-study (Week 104).
Population: as for outcome 1
Measure: Mean (Standard Error); unit: mm/year
Arm/Group | Rosuvastatin 20 mg | Placebo
Number analyzed (Participants) | 272 | 271
mm/year | -0.0011 (0.00191) | 0.0075 (0.00194)
Statistical Analysis 1: Comparison: Rosuvastatin 20 mg vs Placebo; Comparison of annualized rate of change in MeanMean CIMT measurement difference between rosuvastatin 20 mg and placebo; Test type: Other; p = 0.002, Multi-level mixed effects model — Statistical significance of the MeanMean CIMT annualized rate of change between rosuvastatin 20 mg and placebo was evaluated using time-by-treatment interaction term in the model; Estimated mean difference = -0.0086, 95% CI 2-sided [-0.0139 to -0.0032], Standard Error of Mean 0.00272 — [estimate comment as in outcome 1, analysis 1]

6. Secondary Outcome: Percent Change From Baseline in Lipid, Lipoprotein and Apolipoprotein Values at Final Visit: Last Observation Carried Forward (LOCF)
Description: The percent change from baseline at final visit for lipid and lipoprotein measurements (low-density lipoprotein cholesterol [LDL-C], total cholesterol, high-density lipoprotein cholesterol [HDL-C], triglycerides, non-HDL-C, non-HDL-C/HDL-C ratio) and apolipoprotein measurements (apolipoprotein A-I [ApoA-I], apolipoprotein B [ApoB] and ApoB/ApoA-I ratio) was determined by analysis of covariance (ANCOVA) with treatment as a fixed effect and baseline value as a covariate. In the evaluation of change from baseline (Week 0) to the final visit at Week 104, any missing observations were imputed by LOCF.
Time Frame: From baseline (Week 0) to end-of-study (Week 104).
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Rosuvastatin 20 mg | Placebo
Number analyzed (Participants) | 272 | 271
Percent change
  LDL-C: number analyzed (Participants) | 260 | 252
  LDL-C | -26.47 (1.700) | 8.99 (1.727)
  Total Cholesterol: number analyzed (Participants) | 260 | 252
  Total Cholesterol | -20.56 (1.010) | 1.29 (1.026)
  HDL-C: number analyzed (Participants) | 260 | 252
  HDL-C | 5.47 (0.944) | 0.48 (0.959)
  Triglycerides: number analyzed (Participants) | 260 | 252
  Triglycerides | -7.26 (2.575) | 12.38 (2.616)
  Non-HDL-C: number analyzed (Participants) | 260 | 252
  Non-HDL-C | -27.67 (1.344) | 1.82 (1.365)
  Non-HDL-C/HDL-C: number analyzed (Participants) | 260 | 252
  Non-HDL-C/HDL-C | -28.52 (1.637) | 3.23 (1.663)
  ApoB: number analyzed (Participants) | 210 | 214
  ApoB | -24.20 (1.307) | 1.91 (1.295)
  ApoA-I: number analyzed (Participants) | 210 | 214
  ApoA-I | 3.16 (0.784) | 0.96 (0.777)
  ApoB/ApoA-I: number analyzed (Participants) | 210 | 214
  ApoB/ApoA-I | -25.14 (1.450) | 1.63 (1.436)
Statistical Analysis 1: Comparison: Rosuvastatin 20 mg vs Placebo; Treatment difference (rosuvastatin 20 mg - placebo): LDL-C; Test type: Other; p < 0.001, ANCOVA; Least squares mean difference = -35.46, 95% CI 2-sided [-40.23 to -30.70], Standard Error of Mean 2.426 — Treatment as a fixed effect and baseline value as a covariate
Statistical Analysis 2: Comparison: Rosuvastatin 20 mg vs Placebo; Treatment difference (rosuvastatin 20 mg - placebo): total cholesterol; Test type: Other; p < 0.001, ANCOVA; Least squares mean difference = -21.85, 95% CI 2-sided [-24.68 to -19.02], Standard Error of Mean 1.441 — Treatment as a fixed effect and baseline value as a covariate
Statistical Analysis 3: Comparison: Rosuvastatin 20 mg vs Placebo; Treatment difference (rosuvastatin 20 mg - placebo): HDL-C; Test type: Other; p < 0.001, ANCOVA; Least squares mean difference = 5.0, 95% CI 2-sided [2.35 to 7.64], Standard Error of Mean 1.347 — Treatment as a fixed effect and baseline value as a covariate
Statistical Analysis 4: Comparison: Rosuvastatin 20 mg vs Placebo; Treatment difference (rosuvastatin 20 mg - placebo): Triglycerides; Test type: Other; p < 0.001, ANCOVA; Least squares mean difference = -19.65, 95% CI 2-sided [-26.86 to -12.44], Standard Error of Mean 3.671 — Treatment as a fixed effect and baseline value as a covariate
Statistical Analysis 5: Comparison: Rosuvastatin 20 mg vs Placebo; Treatment difference (rosuvastatin 20 mg - placebo): Non-HDL-C; Test type: Other; p < 0.001, ANCOVA; Least squares mean difference = -29.49, 95% CI 2-sided [-33.25 to -25.72], Standard Error of Mean 1.917 — Treatment as a fixed effect and baseline value as a covariate
Statistical Analysis 6: Comparison: Rosuvastatin 20 mg vs Placebo; Treatment difference (rosuvastatin 20 mg - placebo): Non-HDL-C/HDL-C ratio; Test type: Other; p < 0.001, ANCOVA; Least squares mean difference = -31.75, 95% CI 2-sided [-36.33 to -27.16], Standard Error of Mean 2.334 — Treatment as a fixed effect and baseline value as a covariate
Statistical Analysis 7: Comparison: Rosuvastatin 20 mg vs Placebo; Treatment difference (rosuvastatin 20 mg - placebo): ApoB; Test type: Other; p < 0.001, ANCOVA; Least squares mean difference = -26.12, 95% CI 2-sided [-29.73 to -22.50], Standard Error of Mean 1.840 — Treatment as a fixed effect and baseline value as a covariate
Statistical Analysis 8: Comparison: Rosuvastatin 20 mg vs Placebo; Treatment difference (rosuvastatin 20 mg - placebo): ApoA-I; Test type: Other; p = 0.047, ANCOVA; Least squares mean difference = 2.19, 95% CI 2-sided [0.02 to 4.36], Standard Error of Mean 1.104 — Treatment as a fixed effect and baseline value as a covariate
Statistical Analysis 9: Comparison: Rosuvastatin 20 mg vs Placebo; Treatment difference (rosuvastatin 20 mg - placebo): ApoB/ApoA-I ratio; Test type: Other; p < 0.001, ANCOVA; Least squares mean difference = -26.77, 95% CI 2-sided [-30.78 to -22.76], Standard Error of Mean 2.041 — Treatment as a fixed effect and baseline value as a covariate

7. Secondary Outcome: Percent Change From Baseline in Lipid and Lipoprotein Values at Final Visit: Time Weighted Average
Description: The percent change from baseline at final visit for lipid and lipoprotein measurements (LDL-C, total cholesterol, HDL-C, triglycerides, non-HDL-C, non-HDL-C/HDL-C ratio) was determined by ANCOVA with treatment as a fixed effect and baseline value as a covariate. In the evaluation of change from baseline (Week 0), the time-weighted average value was calculated as the value multiplied by the number of days since the last assessment, summed for all observations, and divided by the sum of days between all visits.
Time Frame: From baseline (Week 0) to end-of-study (Week 104).
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Rosuvastatin 20 mg | Placebo
Number analyzed (Participants) | 272 | 271
Percent change
  LDL-C: number analyzed (Participants) | 260 | 252
  LDL-C | -34.89 (1.275) | 4.62 (1.295)
  Total Cholesterol: number analyzed (Participants) | 260 | 252
  Total Cholesterol | -23.98 (0.798) | 1.49 (0.811)
  HDL-C: number analyzed (Participants) | 260 | 252
  HDL-C | 7.07 (0.737) | 3.41 (0.748)
  Triglycerides: number analyzed (Participants) | 260 | 252
  Triglycerides | -9.05 (2.091) | 9.36 (2.124)
  Non-HDL-C: number analyzed (Participants) | 260 | 252
  Non-HDL-C | -32.59 (1.072) | 1.19 (1.089)
  Non-HDL-C/HDL-C: number analyzed (Participants) | 260 | 252
  Non-HDL-C/HDL-C | -34.31 (1.288) | -0.38 (1.308)
Statistical Analysis 1: Comparison: Rosuvastatin 20 mg vs Placebo; Treatment difference (rosuvastatin 20 mg - placebo): LDL-C; Test type: Other; p < 0.001, ANCOVA; Least squares mean difference = -39.51, 95% CI 2-sided [-43.08 to -35.94], Standard Error of Mean 1.819 — Treatment as a fixed effect and baseline value as a covariate
Statistical Analysis 2: Comparison: Rosuvastatin 20 mg vs Placebo; Treatment difference (rosuvastatin 20 mg - placebo): total cholesterol; Test type: Other; p < 0.001, ANCOVA; Least squares mean difference = -25.46, 95% CI 2-sided [-27.70 to -23.23], Standard Error of Mean 1.139 — Treatment as a fixed effect and baseline value as a covariate
Statistical Analysis 3: Comparison: Rosuvastatin 20 mg vs Placebo; Treatment difference (rosuvastatin 20 mg - placebo): HDL-C; Test type: Other; p < 0.001, ANCOVA; Least squares mean difference = 3.67, 95% CI 2-sided [1.60 to 5.73], Standard Error of Mean 1.051 — Treatment as a fixed effect and baseline value as a covariate
Statistical Analysis 4: Comparison: Rosuvastatin 20 mg vs Placebo; Treatment difference (rosuvastatin 20 mg - placebo): Triglycerides; Test type: Other; p < 0.001, ANCOVA; Least squares mean difference = -18.41, 95% CI 2-sided [-24.26 to -12.55], Standard Error of Mean 2.981 — Treatment as a fixed effect and baseline value as a covariate
Statistical Analysis 5: Comparison: Rosuvastatin 20 mg vs Placebo; Treatment difference (rosuvastatin 20 mg - placebo): Non-HDL-C; Test type: Other; p < 0.001, ANCOVA; Least squares mean difference = -33.78, 95% CI 2-sided [-36.78 to -30.78], Standard Error of Mean 1.529 — Treatment as a fixed effect and baseline value as a covariate
Statistical Analysis 6: Comparison: Rosuvastatin 20 mg vs Placebo; Treatment difference (rosuvastatin 20 mg - placebo): Non-HDL-C/HDL-C ratio; Test type: Other; p < 0.001, ANCOVA; Least squares mean difference = -33.93, 95% CI 2-sided [-37.54 to -30.32], Standard Error of Mean 1.836 — Treatment as a fixed effect and baseline value as a covariate

ADVERSE EVENTS:
Time Frame: Treatment Emergent Adverse Events were collected from day of first dose in Week 0 up to and including 10 days following the date of last dose of investigational product or placebo (up to Week 104).
Description: The safety analysis set consisted of all patients who took at least 1 dose of investigational product or placebo. Patients were analyzed according to treatment actually received.
Arm/Group | Rosuvastatin 20 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/272 | 1/268
Serious Adverse Events (participants affected / at risk) | 38/272 | 34/268
Other Adverse Events (participants affected / at risk) | 144/272 | 142/268
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rosuvastatin 20 mg (N=272) | Placebo (N=268)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 2 (2)
Angina unstable (Cardiac disorders) | 0 (0) | 1 (1)
Arrhythmia (Cardiac disorders) | 1 (1) | 1 (1)
Arteriosclerosis coronary artery (Cardiac disorders) | 1 (1) | 2 (2)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1)
Sinus node dysfunction (Cardiac disorders) | 0 (0) | 1 (1)
Vertigo positional (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Goitre (Endocrine disorders) | 1 (1) | 1 (1)
Hyperparathyroidism primary (Endocrine disorders) | 1 (1) | 0 (0)
Thyroid mass (Endocrine disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 2 (3) | 1 (1)
Iridocyclitis (Eye disorders) | 1 (1) | 0 (0)
Pathologic myopia (Eye disorders) | 1 (1) | 0 (0)
Pterygium (Eye disorders) | 0 (0) | 1 (1)
Retinal detachment (Eye disorders) | 1 (1) | 0 (0)
Retinal vein occlusion (Eye disorders) | 0 (0) | 1 (1)
Anal fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 1 (1) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic cyst (Hepatobiliary disorders) | 0 (0) | 1 (1)
Chronic sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Hepatitis viral (Infections and infestations) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Meniscus injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Patella fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pulmonary contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Traumatic fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Investigation (Investigations) | 1 (1) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (4) | 0 (0)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Breast cancer female (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Mycosis fungoides (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Salivary gland cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebral artery stenosis (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 2 (2) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Intercostal neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Hypertonic bladder (Renal and urinary disorders) | 1 (1) | 0 (0)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Henoch-Schonlein purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Arterial thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rosuvastatin 20 mg (N=272) | Placebo (N=268)
Toothache (Gastrointestinal disorders) | 23 (39) | 15 (23)
Nasopharyngitis (Infections and infestations) | 52 (79) | 56 (77)
Upper respiratory tract infection (Infections and infestations) | 49 (74) | 54 (71)
Blood glucose increased (Investigations) | 24 (24) | 18 (18)
Protein urine present (Investigations) | 16 (16) | 9 (10)
Dizziness (Nervous system disorders) | 14 (17) | 16 (24)
Cough (Respiratory, thoracic and mediastinal disorders) | 14 (18) | 15 (19)
Hypertension (Vascular disorders) | 19 (19) | 21 (27)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-03-28): https://cdn.clinicaltrials.gov/large-docs/23/NCT02546323/Prot_000.pdf
  • Statistical Analysis Plan (2019-03-06): https://cdn.clinicaltrials.gov/large-docs/23/NCT02546323/SAP_001.pdf